CLINICAL TRIAL: NCT05447949
Title: Comparison of Dexmedetomidine Versus Dexamethasone as Adjuncts to Levobupivacaine in Ultrasound Guided Erector Spinae Plane Block for Patients Undergoing Modified Radical Mastectomy, Randomized Double-Blinded Comparative Study.
Brief Title: Dexmedetomidine Versus Dexamethasone as Adjuncts in Erector Spinae Plane Block in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohammed Magdy Abdelrahman Elsayed, Assistant Lecturer of Anesthesiology , ICU and Pain Management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MS-536-2021
Record Dates: First submitted 2022-06-27; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Post Operative Pain
Keywords: Modified Radical Mastectomy; Dexmedetomidine; Dexamethasone; Erector Spinae Plane Block; Regional anesthesia
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both the investigator for postoperative pain and the patients will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (ESPB + Dexmedetomidine) (Experimental): Patients received Ultrasound guided ESPB with addition of dexmedetomidine 1 Mcg/kg to 30 ml levobupivacaine 0.25%, N=30 (16)
  Interventions: Procedure: Adjuncts to levobupivacaine in Erector Spinae Plane Block
- Group 2 (ESPB+ dexamethasone) (Experimental): Patients received Ultrasound guided ESPB with addition of dexamethasone 10 mg to 30 ml levobupivacaine 0.25%, N=30 (16)
  Interventions: Procedure: Adjuncts to levobupivacaine in Erector Spinae Plane Block
- Group 3 (ESPB) (Active Comparator): Patients received Ultrasound guided ESPB with 30 ml levobupivacaine 0.25%, N=30
  Interventions: Procedure: Adjuncts to levobupivacaine in Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Adjuncts to levobupivacaine in Erector Spinae Plane Block — The block level will be at T5 with the patient in a sitting position and full aseptic precautions. T5 transverse process; these are recognizable as flat, squared-off acoustic shadows with only a very faint image of the pleura visible. In a longitudinal US view, in which the following layers will be visible superficial to the transverse processes: skin, subcutaneous tissue, trapezius, erector spinae muscle . Skin is topicalized, then echogenic block needle inserted in plane to the ultrasound beam in a cranial-to-caudal direction until contact is made with the T5 transverse process. After aspiration; to avoid intravascular injection, 30 ml of injectate is injected and separation will be seen. 6-13-MHz, linear transducer set for small parts and a depth of 4-6 cm will be used (18-19).

SUMMARY:
The aim of this study is to evaluate the analgesic efficacy and safety of adding dexmedetomidine versus dexamethasone to levobupivacaine in ultrasound guided ESPB for patients undergoing modified radical mastectomy

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy among females. Modified Radical Mastectomy (MRM) is one of the main surgical treatments of breast cancer .The most common modality for anesthesia is general anesthesia with or without regional blocks . Nearly 40-60% of patients undergoing breast surgery experience severe acute postoperative pain, with severe pain persisting for 6-12 months in almost 10-30% of patients (Post Mastectomy Pain Syndrome; PMPS) . This pain can be severe enough to cause long-term disabilities and interfere with sleep and performance of daily activities.

Postoperative pain is usually managed by opioids, yet it is usually associated with side effects including; prolonged sedation, increase in the incidence of recurrence, respiratory depression , nausea , vomiting and ileus. In an attempt to reduce these side effects, thoracic epidural analgesia and paravertebral block became the gold standard regional techniques for breast surgery. However, both techniques may be associated with serious complications such as pneumothorax, spinal cord injury, incompatibility with pre-existing anticoagulation or antiplatelet therapy and hemodynamic instability. Multiple different regional techniques have been developed in the last decade for postoperative pain management of MRM including including erector spinae plane block (ESPB) aiming to be effective and associated with less complications when compared to the gold standard techniques .

ESPB is a simple and safe paraspinal fascial plane block that involves injection of local anesthetic deep in the erector spinae muscle and superficial to the tips of the thoracic transverse processes hoping to block both ventral and dorsal rami of spinal nerves in the paravertebral area. However, regional blocks after a single dose of local anesthetic are of limited duration and efficacy. Hence, the co-administration of adjuvants with local anesthetics may be helpful for prolongation and potentiation of the analgesic effect. Dexmedetomidine is a potent α2agonist of which α2/α1 selectivity is 8 times greater than clonidine and is now emerging as an adjunct to regional and general anesthesia. It can prolong the duration of the nerve block when used with a local anesthetic .Dexamethasone is considered as an adjuvant as it act by reducing the release of inflammatory mediators and by inhibiting discharge of C-fibers. There is a limited number of studies covering the effect of dexmedetomidine versus dexamethasone when added to ESPB, yet they are still lacking in breast surgeries. Our study aims at studying the effect of adding dexmedetomidine compared to dexamethasone as adjuncts to ESPB in modified radical mastectomy.

Objectives:

To identify the intraoperative and postoperative opioid consumption, as well as duration of analgesia and study the effect on hemodynamics.

Hypothesis We hypothesize that the addition of dexmedetomidine to levobupivacaine in US guided ESPB in patients undergoing MRM is superior to either adding dexamethasone to levobupivacaine, or using levobupivacaine alone.

Ethical Considerations The trial will be conducted after approval of departmental and institutional research ethics committee. A written informed consent will be obtained from all participants.

A comparative double-blinded study.

Study setting and location The study will be conducted in the breast operating theatre at National Cancer Institute hospital.

Study population 90 Female patients ASA II,III scheduled for modified radical mastectomy under general anaesthesia.

A. preoperative:

Patient's assessment; History, physical exam, laboratory and radiological investigations at preoperative assessment clinic National Cancer Institute Cairo University. Preoperative assessment on the night of surgery. Patients will be instructed on how to report pain by means of Numeric Pain Rating Scale, in which 0 = "no pain" and 10 = "worst possible pain". An informed consent will be obtained. Preoperative fasting; minimum of 6 hours for food and minimum of 2 hours for water and clear fluids.20G IV cannula is inserted. All patients will be pre-medicated with IV midazolam 0.01-0.02 mg\kg 30 minutes preoperatively. ESPB with either adjuncts or none at all will be done preoperatively with the patients in a lateral position. After allocation of patients to each study group, patients in group 1 will receive dexmedetomidine with levobupivacaine in ESPB, while patients in group 2 will receive dexamethasone with levobupivacaine in ESPB, & patients in group 3 will receive levobupivacaine without adjuncts in ESPB.

Technique of ESPB: The block level will be at T5 with the patient in a lateral position. The ultrasound probe will be placed on the back in a transverse orientation to identify the tip of the T5 transverse process; these are recognizable as flat, squared-off acoustic shadows with only a very faint image of the pleura visible. If the transducer is too lateral, the ribs will be visualized instead; these are recognizable as rounded acoustic shadows with an intervening hyperechoic pleural line. The tip of the transverse process will be centered on the ultrasound screen and the probe will then be rotated into a longitudinal orientation to produce a parasagittal view, in which the following layers will be visible superficial to the acoustic shadows of the transverse processes: skin, subcutaneous tissue, trapezius, erector spinae muscle and T5 transverse process. A skin wheel using 3 ml of lidocaine 1% is made 2-3 cm above the upper aspect of the transducer, then an echogenic block needle will be inserted in plane to the ultrasound beam in a cranial-to-caudal direction until contact is made with the T5 transverse process. Correct location of the needle tip in the fascial plane deep to erector spinae muscle will be confirmed by injecting 0.5-1 ml glucose 5% and seeing the fluid lifting the erector spinae muscle off the transverse process without distending the muscle. After aspiration; to avoid intravascular injection, 30 ml levobupivacaine 0.25% to which dexmedetomidine (1microgram\kg) is added in the first group , while dexamethasone (10 mg) is added to levobupivacaine in the second group, and no adjuncts to levobupivacaine is added to the third group. Upon injection, separation will be seen. 6-13-MHz, linear transducer set for small parts and a depth of 4-6 cm will be used. Fujifilm Sonosite M-Turbo Ultrasound system will be used.

B. Intraoperative:

All patients will be monitored continuously using electrocardiography, non-invasive blood pressure, peripheral oxygen saturation and end tidal carbon dioxide throughout the duration of the surgical procedure. Induction of general anesthesia will be performed using a regimen of IV 2 μg/kg fentanyl and propofol IV 2 mg /kg. Tracheal intubation will be facilitated by using 0.5 mg/kg IV of atracurium. Anesthesia will be maintained with inhaled sevoflurane 2-2.5% in oxygen enriched air (FiO2=0.5). Maintenance doses of atracurium o.1 mg\kg will be provided every 30 minutes. Paracetamol 500 mg and IV ketorolac 30mg will be provided as a part of multimodal analgesia. Rescue analgesia of fentanyl 1 μg/kg will be given if the mean arterial blood pressure or heart rate rises above 20% of the baseline levels. Ringer acetate will be infused to replace the fluid deficit, maintenance and losses, and patients will be mechanically ventilated at an appropriate setting keeping the end-tidal CO2 at 30- 35 mmHg. The first reading of mean arterial pressure (MAP) and heart rate (HR) will be taken before induction of general anesthesia to be defined as a baseline reading, another reading will be taken immediately before surgical incision and at 30-minute intervals intraoperatively. The residual neuromuscular blockade will be reversed using neostigmine (0.05 mg/kg) and atropine (0.02 mg/kg). Extubation will be performed after complete recovery of the airway reflexes.

C. postoperative:

Patients will be transferred to the post-anesthesia care unit (PACU) where the Numeric Pain Rating Scale score, MAP and heart rate will be noted immediately on arrival, then observed for 2 hours & discharged to the ward afterwards. Rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the patient indicates Numeric Pain Rating Scale ≥ 4. The total amount of morphine given in 24 hours will be recorded for the three groups. A maximum dose of 0.5 mg/kg/24hours of morphine is allowed. IV paracetamol 500 mg \6 hours and IV ketorolac 30mg\8 hours will be given as a part of multimodal analgesia. Numeric Pain Rating Scale score, MAP and heart rate will be noted at 4, 8, 12, 16, 20 and 24 hours postoperatively. Side effects such as nausea, vomiting, sedation, respiratory depression (respiratory rate <10/minute) will be recorded. Postoperative nausea and vomiting (PONV), will be rated on a four-point verbal scale; (none =no nausea, mild =nausea but no vomiting, moderate=vomiting one attack, severe =vomiting >one attack). 0.1 mg/kg of IV ondansetron will be given to patients with moderate or severe postoperative nausea and vomiting . Sedation will be assessed in the PACU with Ramsay scores.(1 = anxious or restless or both; 2 = cooperative, orientated, and tranquil; 3= responding to commands; 4 = brisk response to stimulus; 5 = sluggish response to stimulus; and 6 = no response to stimulus). A Ramsay score of 5 or 6 will be considered excessively high sedation levels; a Ramsay score of 2 to 4 will be considered adequate sedation levels needing observation; a Ramsay score of 1 will be considered inadequate or insufficient sedation levels .

Sample size As there was no study reporting results on a similar hypothesis, sample size was calculated based on the results of pilot study;SPSS version 23.0 was used to generate a list of 20 subjects who were randomly assigned into two groups each of 10 for the following treatment A) ESPB + Dexamethasone B) ESPB + Precedex Assuming a pooled standard deviation of 2.37 units, the study would require a sample size of thirty for each group (i.e. a total sample size of 60, assuming equal group sizes), to achieve a power of 90% and a level of significance of 1% (two sided), for detecting a true difference in means of post operative morphia consumption between ESPB + Dexamethasone and ESPB + Precedex groups of -2.4 (i.e. 2.4 - 4.8) units.

Statistical analysis PSS version 27.0 will be used in data analysis. Quantitative variables were tested for normality to select appropriate statistical tests. Mean and standard deviation described quantitative data with median and range. Comparison of means (or medians) of two independent groups will be done using t test. To show the effect of time on vitals, parametric repeated measures ANOVA or Friedman test will be used to show changes overtime both intra and post-operative. Post-hoc test will be used for pairwise comparisons and will be Tucky adjusted. Chi-square and Fisher Exact were used for testing proportion independence. P value was always two tailed and set significant at 0.05 level

ELIGIBILITY:
Inclusion Criteria:

* Type of surgery; Modified Radical Mastectomy (MRM)
* Physical status ASA II, III.
* Age ≥ 18 and ≤ 65 Years.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* Patient's refusal
* Age <18 years or >65 years
* BMI <20 kg/m2 and >35 kg/m2
* Known sensitivity or contraindication to drug used in the study (local anaesthetics, opioids).
* History of psychological disorders and/or chronic pain.
* Contraindication to regional anaesthesia e.g. local sepsis, pre- existing peripheral neuropathies and coagulopathy.
* Severe respiratory or cardiac disorders.
* Advanced liver or kidney disease. Pregnancy.
* Physical status ASA IV.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Total amount of morphine consumed postoperatively for 24 hours. | 24 hours
  Total amount of morphine consumed postoperatively in mg for 24 hours.

SECONDARY OUTCOMES:
Total amount of fentanyl consumed intraoperatively. | Duration of surgery
  Total amount of fentanyl in Mcg consumed intraoperatively.
Change in heart rate intraoperatively | Duration of surgery
  Intraoperative measurement of HR at 30 minutes interval in comparison to baseline reading.
Change in mean arterial blood pressure intraoperatively | Duration of surgery
  Intraoperative measurement of MAP at 30 minutes interval in comparison to baseline reading.
Postoperative sedation according to Ramsay scores. | 24 hours
  Scores at 0,2,4,8,12,16,20,24 hours. (1 = anxious or restless or both; 2 = cooperative, orientated, and tranquil; 3= responding to commands; 4 = brisk response to stimulus; 5 = sluggish response to stimulus; and 6 = no response to stimulus). A Ramsay score of 5 or 6 will be considered excessively high sedation levels; a Ramsay score of 2 to 4 will be considered adequate sedation levels needing observation; a Ramsay score of 1 will be considered inadequate or insufficient sedation levels (21).
Time to first rescue analgesia. | 24 hours
  Duration of analgesic effect until the time of 1st rescue analgesia
Numeric Pain Rating Scale score, both at rest and during movement | 24 hours postoperative
  Scores will be recorded in the PACU, and every 4 hours until 24 hours postoperatively.
  Patients will be instructed on how to report pain by means of Numeric Pain Rating Scale, in which 0 = "no pain" and 10 = "worst possible pain".
Block related complications | 24 hours postoperative
  Complications related to the block such as local anaesthetic systemic toxicity and vascular injury.
Patient's satisfaction | 24 hours postoperative
  the patient will be classified in this group to satisfied or not.
Incidence of Postoperative nausea and vomiting (PONV). | 24 hours postoperative
  PONV will be rated on a four-point verbal scale; (none =no nausea, mild =nausea but no vomiting, moderate=vomiting one attack, severe =vomiting >one attack). 0.1 mg/kg of IV ondansetron will be given to patients with moderate or severe postoperative nausea and vomiting (20).

CONTACTS AND LOCATIONS:
Overall Officials: Ashgan R Ali, Professor, Study Chair — Anaesthesiology Faculty of Medicine - Cairo University; Heba I Ahmed, Ass. Professor, Study Director — Anaesthesiology Faculty of Medicine - Cairo University; Reham M Gamal, Lecturer, Study Director — Anaesthesiology National Cancer Institute - Cairo University; Mohammed M Abdelrahman, Ass. Lecturer, Study Director — Anaesthesiology National Cancer Institute - Cairo University; Norhan H El Emam, Resident, Principal Investigator — Anaesthesiology National Cancer Institute - Cairo University
Locations (1):
- National Cancer Institute - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No